CLINICAL TRIAL: NCT00214058
Title: Phase II Evaluation of Weekly Docetaxel in Combination With Weekly Carboplatin in the Treatment of Recurrent Epithelial Ovarian Carcinoma
Brief Title: Weekly Carboplatin/Docetaxel for Recurrent Ovarian/Peritoneal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Aventis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CO02701; 2002-224 (Other: Institutional Review Board); A532820 (Other: UW Madison); SMPH/OBSTET & GYNECOL (Other: UW Madison)
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2019-11-19 (Actual); Status verified 2008-06

CONDITIONS: Ovarian Carcinoma; Primary Peritoneal Carcinoma
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Carboplatin; Docetaxel

INTERVENTIONS:
Drug: Carboplatin
Drug: Docetaxel

SUMMARY:
The purpose of this study is to determine the safety and efficacy of this regimen in women with ovarian or peritoneal cancer

ELIGIBILITY:
Inclusion Criteria:

* Recurrent ovarian or peritoneal cancer

Exclusion Criteria:

* No prior chemotherapy

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Enrollment: 36
Dates: Start 2002-08; Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
Safety and Efficacy

SECONDARY OUTCOMES:
QOL

CONTACTS AND LOCATIONS:
Overall Officials: David M Kushner, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Hospital and Clinics, Madison, Wisconsin, United States

REFERENCES:
- See also: University of Wisconsin Carbone Cancer Center — https://cancer.wisc.edu